CLINICAL TRIAL: NCT00182806
Title: Phase II Study of Irinotecan Followed by Gemcitabine in NSCLC Following Failure of Platinum Based Therapy
Brief Title: Irinotecan and Gemcitabine in Treating Patients With Recurrent or Progressive Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000441226; RPCI-I-31204
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gemcitabine hydrochloride — IV over 30 minutes on days 2 and 9. Courses repeat every 21 days.
Drug: irinotecan hydrochloride — IV over 90 minutes on days 1 and 8. Courses repeat every 21 days.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Irinotecan may also increase the effectiveness of gemcitabine. Giving irinotecan together with gemcitabine may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving irinotecan together with gemcitabine works in treating patients with recurrent or progressive stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate (complete and partial response) in patients with recurrent or progressive stage IIIA-IV non-small cell lung cancer treated with irinotecan and gemcitabine.

Secondary

* Determine the median time to progression in patients treated with this regimen.

OUTLINE: This a non-randomized, open-label, multicenter study.

Patients receive irinotecan IV over 90 minutes on days 1 and 8 and gemcitabine IV over 30 minutes on days 2 and 9. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 1 month and then every 8 weeks thereafter.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 16 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC), meeting 1 of the following stage criteria:

  * Stage IIIA or IIIB disease

    * Progressive disease
  * Stage IV disease

    * Failed 1 prior platinum-based chemotherapy regimen, including adjuvant therapy
* Measurable or evaluable disease, as defined by 1 of the following criteria:

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR > 10 mm by spiral CT scan
  * Lesions apparent on CT scan that do not meet the criterion for measurability
* Brain metastases allowed provided patient has received definitive therapy for metastases, is asymptomatic, and has extra-CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* More than 12 weeks

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* AST and ALT ≤ 1.5 times normal
* Alkaline phosphatase < 1.5 times normal
* Bilirubin ≤ 1.3 mg/dL

Renal

* Creatinine ≤ 1.6 mg/dL OR
* Creatinine clearance ≥ 50 mL/min

Cardiovascular

* No unstable angina
* No congestive heart failure
* No myocardial infarction within the past 3 months
* No life-threatening ventricular arrhythmia requiring maintenance therapy

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after completion of study treatment
* No uncontrolled seizure disorder
* No uncontrolled diabetes mellitus
* No active infection requiring systemic therapy
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No other unstable or serious condition

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy
* Prior irinotecan allowed
* No prior gemcitabine
* No more than 1 prior chemotherapy regimen for NSCLC, excluding gefitinib
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* Not specified

Other

* More than 1 month since prior participation in another clinical trial using an investigational agent
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2004-09; Primary Completion 2007-09 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Objective response (complete, partial, and stable disease)

SECONDARY OUTCOMES:
Median time to progression

CONTACTS AND LOCATIONS:
Overall Officials: Nithya Ramnath, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Result] Ramnath N, Yu J, Khushalani NI, Gottlieb RH, Schwarz JK, Iyer RV, Rustum YM, Creaven PJ. Scheduled administration of low dose irinotecan before gemcitabine in the second line therapy of non-small cell lung cancer: a phase II study. Anticancer Drugs. 2008 Aug;19(7):749-52. doi: 10.1097/CAD.0b013e328301c54f. PMID 18594219